CLINICAL TRIAL: NCT01467167
Title: Utility of the Smart Pilot View in Clinical Practice: A Two Center Prospective Observational Study
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: SPV_Utility_V7
Record Dates: First submitted 2011-09-14; First posted 2011-11-08 (Estimated); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia,General
Keywords: Anesthesia; Smart Pilot View; Pain control; Recovery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Baseline: Baseline group in which patients are anesthetized without the use of Smart Pilot View, according to common practice.
- Smart Pilot View Group: Study group in which patients are anesthetized with the use of Smart Pilot View.

SUMMARY:
Recently, a new software program for anesthesia has been developed, called Smart Pilot View. This program monitors the patient, the anesthetic drugs given, and the calculated depth of the anesthesia. The purpose of this study is to determine whether the use of this program improves the quality of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* General anesthesia
* American Society of Anesthesiologists Physical Status: I - III
* Age 18 to 90 years

Exclusion Criteria:

* Combined regional and general anesthesia
* Expected surgery duration < 30 minutes
* Central nervous system (CNS) diseases (dementia, cerebrovascular accident, seizures, psychiatric diseases)
* Regular intake of CNS active drugs (benzodiazepines, antidepressants, antipsychotics, anticonvulsants)
* Heart surgery on cardio-pulmonary bypass
* Relevant hepatic disease (Child B or higher)
* BMI >35
* Overt signs of alcohol abuse
* Contraindications or allergies to drugs used in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery under general anesthesia scheduled for neurosurgery, gynecology and ear nose and throat surgery.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Anesthesia Quality Score | up to 1 week From start of induction until discharge from post-anesthesia care unit (PACU)
  Anesthesia Quality Score (AQS) is defined as the percentage of time the BIS is within the range of 40-60 AND the mean arterial pressure is within the range of 60-80 mmHg.

SECONDARY OUTCOMES:
Total anesthetic drug doses | up to 1 week From start of induction until discharge from post-anesthesia care unit (PACU)
Mean intra-operative Noxious Stimulation Response Index (NSRI) | 1 day During surgery (until skin closure)
  The Noxious Stimulation Response Index (NSRI) is based on a hierarchical interaction propofol-remifentanil model. With this model, the predicted propofol and remifentanyl concentrations can make a prediction about a respons to a certain stimulus, such as shaking and shouting, or a noxious stimulus.
Number of doses of vasoactive substances | up to 1 week From start of induction until discharge from post-anesthesia care unit (PACU)
  The number of doses of vasoactive substances given to maintain an adequate perfusion pressure.
Number of events with motor and vegetative (tearing, sweating) responses | up to 1 week From start of induction until discharge from post-anesthesia care unit
  The total number of events in which the patient displays vegetative reactions such as tearing and sweating, in respons to a noxious stimulus during surgery.
Recovery times (skin closure to extubation; skin closure to orientation) | up to 1 week From end of surgery (skin closure) until discharge from post-anesthesia care unit (PACU)
  The time it takes for the patient to recover from anesthesia: the time from skin closure until the patient is sufficiently awake to be extubated, and the time from skin closure until full orientation of the patient.
Early postoperative pain control measured by visual analog scale and total morphine dose | up to 1 day From end of surgery (skin closure) until discharge from post-anesthesia care unit (PACU)
  Assess the adequacy of pain control during the early postoperative stage, measured by the visual analog scale and the total dose of morphine immediately postoperatively and during PACU stay.
Workload of anesthesist, measured by the NASA Taskload Index | up to 1 day From start of induction until transportation to PACU
  Assess the workload the anesthetist experiences while working with the Smart Pilot View

CONTACTS AND LOCATIONS:
Locations (2):
- University Medical Center Groningen (UMCG), Groningen, Netherlands
- University Hospital of Bern, Bern, Switzerland

REFERENCES:
- [Derived] Kuizenga MH, Vereecke HEM, Absalom AR, Bucher CH, Hannivoort LN, van den Berg JP, Schmalz L, Struys MMRF, Luginbuhl M. Utility of the SmartPilot(R) View advisory screen to improve anaesthetic drug titration and postoperative outcomes in clinical practice: a two-centre prospective observational trial. Br J Anaesth. 2022 Jun;128(6):959-970. doi: 10.1016/j.bja.2022.02.033. Epub 2022 Mar 28. PMID 35361490